CLINICAL TRIAL: NCT07294105
Title: Investigation of the Relationship Between Periodontal Disease and Serum and Gingival Crevicular Fluid Sclerostin and Tumor Necrosis Factor- α Levels in Women With Postmenopausal Osteoporosis
Brief Title: Relationship Between Periodontal Disease and Postmenopausal Osteoporosis
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Mujde Cilkus, Research Assistant, Recep Tayyip Erdogan University
Other Study IDs: RecepTayyipErdoganU-DHF-MC-01
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Disease; Postmenopausal Osteoporosis (PMO)
Keywords: Periodontitis; Postmenopausal osteoporosis; Sclerostin; Tumor necrosis factor
MeSH Terms: conditions — Periodontal Diseases; Osteoporosis, Postmenopausal; Periodontitis; Sclerosteosis | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid (GCF) samples will be collected and stored at -80°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group C (Control): Periodontally and systemically healthy women without osteoporosis (n=20)
  Interventions: Other: clinical assessment; Diagnostic Test: Radiographic Evaluation
- Group P (Experimental): Women with periodontitis and without osteoporosis (n=20)
  Interventions: Other: clinical assessment; Diagnostic Test: Radiographic Evaluation
- Group O (Experimental): Periodontally healthy women with osteoporosis (n = 20)
  Interventions: Other: clinical assessment; Diagnostic Test: Radiographic Evaluation
- Group OP (Experimental): Women with periodontitis and osteoporosis (n = 20)
  Interventions: Other: clinical assessment; Diagnostic Test: Radiographic Evaluation

INTERVENTIONS:
Other: clinical assessment — The plaque index (PI) is a quantitative measure used to evaluate the presence and amount of dental plaque on tooth surfaces. Her dişin dört yüzeyi incelenir ve plak varlığına göre 0'dan 3'e kadar puanlanır.
  Other Names: Clinical Index and Measurements
Diagnostic Test: Radiographic Evaluation — Bone Mineral Density measurements will perform using the Stratos dR 2D Fan Beam DXA device. L1-L4, femoral neck, and femur total T-score values, as well as BMD (gr/cm3) values, will record for all patients.
  Other Names: Bone Mineral Density Measurements
Other: clinical assessment — The gingival index (GI) is a clinical parameter that evaluates the degree of gingival inflammation by examining changes in color, texture, and bleeding tendency of the gingiva. Her dişin dört yüzeyi incelenir ve diş eti rengi, ödemi ve kanama durumuna göre 0'dan 3'e kadar puanlanır.
  Other Names: klinik indeksler ve ölçüm
Other: clinical assessment — Sondlamada kanama indeksi diş etlerinin sondlama (periodontal prob ile hafif dokunma) veya fırçalama sonrası kanama eğilimini ölçer. Diş eti dokusundaki inflamasyonun derecesi hakkında bilgi verir. Ainamo & Bay (1975) - Bleeding on Probing (BOP) Index Periodontal sondun dişeti oluğuna yerleştirilmesinden 10-15 saniye sonra kanama olup olmadığı gözlenir.
  Other Names: klinik indeksler ve ölçüm
Other: clinical assessment — Probing Pocket Depth (PPD), diş ile diş eti arasındaki boşluğun (gingival sulkus veya periodontal cep) diş eti kenarından (gingival margin) cep tabanına (junctional epithelium) kadar olan dikey mesafesidir.
  Bu ölçüm, periodontal sond (genellikle milimetrik işaretlere sahip ince metal bir alet) ile yapılır.
  Other Names: klinik indeksler ve ölçümler
Other: clinical assessment — Clinical attachment level measurement diş eti kenarından (gingival margin) değil, mine-sement sınırı (cementoenamel junction - CEJ) ile cep tabanı (junctional epithelium) arasındaki dikey mesafedir.
  Bu ölçüm, periodontal destek dokularının kalıcı kaybını gösterir.
  Other Names: klinik indeksler ve ölçümler

SUMMARY:
Elevated sclerostin levels in serum and alveolar bone of osteoporotic patients may exert deleterious effects on the periodontium, thereby contributing to the progression and increased severity of periodontal disease. Moreover, sclerostin is considered a potential biomarker for elucidating the shared pathophysiological mechanisms linking postmenopausal osteoporosis and periodontitis

DETAILED DESCRIPTION:
In this study, it has aimed to reveal the relationship between postmenopausal osteoporosis and periodontitis by comparing inflammatory (TNF-α) and bone destruction biomarker (sclerostin) levels in serum and GCF and clinical periodontal parameters in postmenopausal women with decreased BMD. A total of 80 postmenopausal female have included in our study. Patients have divided into 4 groups according to radiological and clinical examination results as control (Group K), periodontitis (Group P), osteoporosis (Group O) and osteoporosis-periodontitis (Group OP). Clinically, PI, GI, BI, PPD and CAL have measured. TNF-α and sclerostin levels have measured by ELISA method in serum and DOS samples. In addition, L1-L4, femoral total and femoral neck BMD values have determined by DXA method. For statistical analyses, Shapiro Wilk test, Mann Whitney U test, Anova test, Kruskal Wallis test, Post Hoc Bonferroni test, Pearson Chi-Square test, Fisher's Exact test, Pearson and Spearman correlation have used. Results: Serum sclerostin level of Group OP and Group P and GCF sclerostin level of Group OP, Group P and Group O have higher than Group K (p<0.05). A positive correlation has found between serum sclerostin level and serum TNF-α (p=0.013, r=0.278) with GCF TNF-α (p=0.001, r=0.356) levels (p<0.05). A positive correlation has found between GCF TNF-α (p=0.002, r=0.334) and GCF sclerostin level (p<0.05).

The increased level of sclerostin in serum and GCF in osteoporosis patients may increase the severity of periodontal disease by creating a destructive effect on the periodontium; It is also thought that it can be used as a biomarker to elucidate the common mechanism in the relationship between postmenopausal osteoporosis and periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 40 years and older in the postmenopausal period,
* Individuals diagnosed with osteoporosis or healthy individuals without osteoporosis, as determined by DXA testing of the hip or spine,
* Individuals who had been postmenopausal for ≥6 months and had not received hormone replacement therapy,
* Patients who did not smoke or consume alcohol,
* Female patients who were periodontally healthy or diagnosed with Stage 2-3, Grade A periodontitis

Exclusion Criteria:

* Patients with chronic renal and hepatic insufficiency; malignant diseases such as diabetes mellitus, leukemia, multiple myeloma, and widespread carcinoma; chronic inflammatory rheumatic diseases such as rheumatoid arthritis and ankylosing spondylitis; and those using drugs that may affect bone metabolism (glucocorticoids, heparin, methotrexate, anticonvulsants),
* Those who had received antibiotic therapy in the previous 3 months or any medication for osteoporosis treatment,
* Patients who had undergone surgical or non-surgical periodontal treatment within the previous 6 months,
* Patients who did not wish to continue participation in the study at the midpoint or at the end of the study.

Ages: 43 Years to 78 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Postmenopausal female patients applying to the Periodontics Clinic of Recep Tayyip Erdoğan University Faculty of Dentistry
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Serum Sample Collection | 6 month
  Venous blood samples will from the left antecubital fossa of the patients
Collection and Quantification of Gingival Crevicular Fluid Samples | 6 month
  Based on the patient's clinical examination status 24 hours after the periodontal clinical measurements, the deepest probable pocket area for individuals with periodontitis, each in six separate quadrants, will sellect for GCF samples. For periodontally healthy individuals, four teeth with a pocket depth of <3 mm, a gingival and plaque index of 0, and no bleeding were selected.

CONTACTS AND LOCATIONS:
Overall Officials: MUJDE CİLKUS, Research Assistant, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdoğan University, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No